CLINICAL TRIAL: NCT05131711
Title: Combination of Stereotactic Radiosurgery and Enhanced Immunotherapy for Recurrent Glioblastomas (inSituVac2)(CSREIG)
Brief Title: Combination of Stereotactic Radiosurgery and Enhanced Immunotherapy for Recurrent Glioblastomas(inSituVac2)(CSREIG)
Acronym: CSREIG
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Song Lin, Neurosurgery, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B0012
Record Dates: First submitted 2021-11-16; First posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Glioblastoma
Keywords: recurrent glioblastomas; stereotactic radiosurgery; enhanced immunotherapy
MeSH Terms: conditions — Glioblastoma | interventions — Radiosurgery; Granulocyte-Macrophage Colony-Stimulating Factor; streptococcal preparation 722; manganese chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rGBM Group with combined stereotactic radiosurgery and enhanced immunotherapy (Experimental): Patients with rGBMs will receive combined stereotactic radiosurgery and enhanced immunal adjuvants (GM-CSF, Sapylin, MnCl2). The safety and efficacy will be analyzed.
  Interventions: Combination Product: Combined stereotactic radiosurgery and enhanced immunotherapy
- rGBM Group with (No Intervention): After biopsy or tumor resection, this rGBM group was treated with FDA-approved strategies proposed by the MDT group.

INTERVENTIONS:
Combination Product: Combined stereotactic radiosurgery and enhanced immunotherapy — Patients will be administrated immunal adjuvants intratumorally and systemically with concurrent stereotactic radiosurgery.
  Other Names: stereotactic radiosurgery and GM-CSF, Sapylin, MnCl2
  Arms: rGBM Group with combined stereotactic radiosurgery and enhanced immunotherapy

SUMMARY:
The study will investigate combined stereotactic radiosurgery and enhanced immunotherapy for recurrent glioblastomas. Immune adjuvants will be injected intratumorally and systemically to induce antitumor-specific immunity after radiation induced immunological tumor cell death (ICD). With radiation, tumor cells release tumor antigens that are captured by antigen presenting dendritic cells. Immune adjuvants promote the presentation of tumor antigens and the priming of antitumor T lymphocytes. The combined treatment induces and amplifies the specific antitumor immunity in patients with recurrent glioblastomas, prolonging survivals of patients.

DETAILED DESCRIPTION:
Recurrent glioblatoma (rGBM) is an aggressive malignancy with a poor prognosis. There is no standard therapy and survival is less than 9 months. Recently, personalized cancer immunotherapy has shown great promise in treating different types of cancers. However, effective immunotherapies for rGBMs have yet to be established. The last clinical trial (inSituVac1) showed promised results and this study was based on it. We will investigate whether combining stereotactic radiosurgery with intratumoral and systemic administration of enhanced immune adjuvants will improve the treatment outcome of rGBMs. We will use several immune adjuvants that activate innate and adaptive immunity.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed rGBM
* 2. Age18-65
* 3. Participants had undergone maximal surgical resection
* 4. Amount of dexamethasone was not more than 2mg/ days
* 5. Ability and willingness to sign informed consent
* 6. Karnofsky Performance Score of 70 or more
* 7. Normal liver and kidney function
* 8. Not accepted other treatment plan during the immunotherapy

Exclusion Criteria:

* 1. Not conforming to the standard
* 2. Systemic illness or medical condition may pose additional risk,including cardiac, incompensated renal or liver function abnormalities;inflammatory and immune system diseases of rheumatic arthritis
* 3. Received other drugs for glioma therapy 60 days before participated
* 4. Allergy to immune adjuvant
* 5. Nervous system disease and diffuse leptomeningeal disease
* 6. Amount of dexamethasone was more than 2mg/days during the immunotherapy
* 7. Pregnant or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-11-16 (Estimated); Study Completion 2023-11-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 2 years
  Adverse events during and after the combined treatment
Progression-free Survival | 2 years
  Disease progression free survival time after combined treatment

SECONDARY OUTCOMES:
overall survival | 2 years
  Overall survival time after the combined treatment

CONTACTS AND LOCATIONS:
Overall Officials: Song Lin, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No